CLINICAL TRIAL: NCT04743206
Title: Airway Clearance for Pediatric and Adult Cystic Fibrosis Patients Using a Portable Intra-Pulmonary Percussion Device (PIAPD)
Brief Title: Airway Clearance for Pediatric and Adult Cystic Fibrosis Patients Using a Portable Intra-Pulmonary Percussion Device
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: recruitment difficulty due to COVID recruitment difficulty due to covid
Sponsor: University of Florida (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: IRB201902662; OCR39724 (Other: UF Oncore)
Record Dates: First submitted 2021-02-03; First posted 2021-02-08 (Actual); Results first posted 2024-11-19 (Actual); Last update posted 2024-11-19 (Actual); Status verified 2024-10

CONDITIONS: Cystic Fibrosis
Keywords: Airway Clearance
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Intervention Model Description: This is a pilot study where the investigators aim to compare initial use of the standard airway clearance device (SACD) with subsequent use of a PIAPD in patients with stable cystic fibrosis ages 6 -21 years. The primary hypothesis (Stated as Null) being that there is no effect of PIAPD on FEV1 2 hours after use, there is no effect on perception of effort and efficacy for the PIAPD.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- PIAPD-Portable Internal Airway Percussion device (Experimental): There will be an outpatient arm using the PIAPD-Portable Internal Airway Percussion Device.
  Interventions: Device: Portable Internal Airway Percussion device
- SACD-Standard Airway Clearance device (Active Comparator): There will be an Outpatient Arm using the SACD, VEST (High Frequency Chest Wall Oscillation VEST) Standard Airway Clearance Device.
  Interventions: Device: Standard Airway Clearance device

INTERVENTIONS:
Device: Standard Airway Clearance device — Subjects will be using their home standard airway clearance device, VEST (High Frequency Chest Wall Oscillation VEST) for 2 weeks followed by PIAPD.
  Arms: SACD-Standard Airway Clearance device
Device: Portable Internal Airway Percussion device — Subjects will be using the investigational device, PIAPD (Portable Internal Airway Percussion Device) for 2 weeks.
  Arms: PIAPD-Portable Internal Airway Percussion device

SUMMARY:
This is a pilot study where the investigators aim to compare initial use of the standard airway clearance device (SACD), most commonly used being High frequency vest airway clearance system (VEST) with subsequent use of a Portable Intra-Pulmonary Percussion Device (PIAPD) in patients with cystic fibrosis (CF) ages 6 -21 years. The primary hypothesis is that there is no effect of PIAPD on Forced expiratory volume in 1 second (FEV1) 2 hours after use, there is no effect on perception of effort and efficacy for the PIAPD. If both are equally effective, the latter device provides an alternative that is both cheaper and portable.

ELIGIBILITY:
Inclusion Criteria:

* Ages 6-21 years
* Cystic fibrosis stable by physician assessment
* Assents to forego additional experimental treatments during the study
* Currently using and familiar with airway clearance therapy for treatment of cystic fibrosis
* Participant (or parent or legal guardian if the participant is a minor) is willing to provide -----Informed Consent

Exclusion Criteria:

* FEV1 < 40% predictive
* Pneumothorax
* Hemoptysis
* Coronavirus disease (COVID) 19 diagnosis within last 14 days
* Any condition that, in the opinion of the investigator, would interfere with the study conduct or the safety of the participant

  * Additional Exclusion Criteria: Outpatient Arm (in addition to general exclusion criteria above) Decrease in FEV1 > 10% from baseline over last 12 months Antibiotic Initiation for acute CF exacerbation Hospitalization for CF Exacerbation
  * Additional Exclusion Criteria: Inpatient Arm (in addition to general exclusion criteria above) Failure to increase FEV1 > 10 % from initial Pulmonary function testing (PFTs) on admission by day 9 of hospitalization.

Ages: 6 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 1 (Actual)
Dates: Start 2021-05-18 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-08-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Silvia Delgado Villalta, MD, Principal Investigator — University of Florida
Locations (1):
- UF Medical Plaza Pulmonary Clinic, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Only one patient was recruited to the study. The patient was outpatient. There were difficulties with recruitment related to COVID-19 pandemic, difficulties obtaining pulmonary function testing related to Covid-19 pandemic, limited staff.
Groups:
- SOC Airway Clearance Device (VEST) Followed by PIAPD-Portable Internal Airway Percussion Device: Subjects will use Standard of Care (SCA) airway clearance Device (VEST) for 2 weeks followed by Interventional Airway Clearance Device (PIAPD) for 2 weeks.
  Forced Expiratory Volume in 1 Second (FEV1) will be measured by Smart One® portable home spirometer.
Period: SOC Airway Clearance Device ( VEST)
Arm/Group | SOC Airway Clearance Device (VEST) Followed by PIAPD-Portable Internal Airway Percussion Device
Started | 1
Completed | 1
Not Completed | 0
Period: PIAPD
Arm/Group | SOC Airway Clearance Device (VEST) Followed by PIAPD-Portable Internal Airway Percussion Device
Started | 1
Completed | 1
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: only one patient was recruited. The patient participated as outpatient.
Groups:
- SACD-Standard Airway Clearance Device Followed by PIAPD: There will be an Outpatient Arm using the SACD for 2 weeks followed by PIAPD for 2 weeks.
Arm/Group | SACD-Standard Airway Clearance Device Followed by PIAPD
Number analyzed (Participants) | 1
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 1
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 1
  Male | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 1
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 1

OUTCOME MEASURES:

1. Primary Outcome: Oxygen Saturation % by Pulse Oximetry
Description: oxygen saturation will be obtained by home pulse oximeter device.
Time Frame: O2 saturation measured immediately prior to treatment and 2 hours after treatment - one-time pre/post treatment in week 1; and one-time pre/post treatment in week 2
Measure: Number; unit: percentage of oxygen saturated hemoglobi
Groups:
- SOC Airway Clearance Device (VEST) Followed by PIAPD-Portable Internal Airway Percussion Device: Subjects will use Standard of Care (SCA) airway clearance Device (VEST) for 2 weeks followed by Interventional Airway Clearance Device (PIAPD) for 2 weeks.
Arm/Group | SOC Airway Clearance Device (VEST) Followed by PIAPD-Portable Internal Airway Percussion Device
Number analyzed (Participants) | 1
percentage of oxygen saturated hemoglobi
  week 1 Vest pretreatment | 98
  week 1 Vest post treatment | 98
  week 2 Vest pretreatment | 97
  week 2 Vest post treatment | 98
  week 1 PIAPD pretreatment | 98
  week 1 PIAPD post treatment | 98
  week 2 PIAPD pretreatment | 99
  week 2 PIAPD post treatment | 98

ADVERSE EVENTS:
Time Frame: The collection time was between June 17, 2021 to June 26, 2021 - please clarify this is a 4 week study
Description: NO Adverse events reported
Groups:
- Vest Followed by PIADD: Vest airway clearance treatment for 2 weeks, followed by PIADD airway clearance treatment for 2 weeks
Arm/Group | Vest Followed by PIADD
All-Cause Mortality (participants affected / at risk) | 0/1
Serious Adverse Events (participants affected / at risk) | 0/1
Other Adverse Events (participants affected / at risk) | 0/1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2021-03-09): https://cdn.clinicaltrials.gov/large-docs/06/NCT04743206/Prot_SAP_001.pdf